CLINICAL TRIAL: NCT05435976
Title: Safety and Clinical Performance of a Non-cross-linked Porcine Acellular Dermal Matrix Used in Dental Surgery
Brief Title: Evaluation of a Non-cross-linked Porcine Acellular Dermal Matrix Used in Dental Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Meccellis Biotech (Industry)
Responsible Party: Sponsor
Other Study IDs: DS_01_CIP
Record Dates: First submitted 2022-06-22; First posted 2022-06-28 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Dental Surgery
Keywords: dental regeneration of soft tissue; biological mesh

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: CELLIS Dental (Porcine Acellular Dermal Matrix, PADM) — Biological membranes used in dental surgery

SUMMARY:
The general objective of the study is to confirm the medium/long-term safety and clinical performance of the CELLIS Dental membrane used in dental surgery and to identify emerging risks in comparison to clinical data related to other treatment modalities.

The present study will be a prospective multicentric non-randomized and noncontrolled trial involving 50 patients followed for 24 months. The study will be conducted in France in 4 investigational centres.

DETAILED DESCRIPTION:
The study will be prospective, multicentric, single-arm observational (non-interventional) to evaluate the safety and performance of the CELLIS Dental membrane used in dental surgery.

All evaluations will be performed and products used according to the usual practice and the device IFU. CELLIS Dental will be used in accordance with its approved labelling.

The study will be conducted in France in 4 investigational centres including 50 patients scheduled for dental regeneration of soft tissue defects and development of soft tissues around teeth or implants.

Each patient will participate in one assessment period including a preoperative visit followed by the surgical procedure.

Patients will return for ambulatory visits on day 15 (+/- 5 days), on month 3 (+/- 2 weeks), on month 12 (+/- 2 weeks) and on month 24 (+/-2 weeks) post-surgery.

CELLIS Dental will be implanted following standard techniques according to indications:

* Treatment of recession defects (gingival recession),
* Soft tissue augmentation around teeth and implants,
* Soft tissue grafting in combination with GBR/GTR,
* Covering/sealing of extraction sockets.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥18 years,
* Patient with an indication of keratinized soft tissue regeneration in the buccal cavity and/or keratinized soft tissue development around teeth or implants,
* Patient being informed of his participation to the study and of the follow-up visits, and having given his written informed consent,
* Patient being informed of the porcine origin of the device in advance of the procedure.

Exclusion Criteria:

* Patient with known hypersensitivity to porcine materials,
* Patient with acute or chronic infection or inflammation of the buccal cavity,
* Patient with a general illness contra-indicated for implantology, periodontology, stomatology, cranio-maxillo-facial surgery,
* Patient who is pregnant,
* Patient who is incapacitated including protected and deprived of liberty person,
* Patient having refused to participate in the study,
* Patient refusing to return for the follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult with an indication of keratinized soft tissue regeneration in the buccal cavity and/or keratinized soft tissue development around teeth or implants
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of adverse events including reoperation following a complication and matrix removal | From the surgical procedure throughout the entire 24-month follow-up period
  Percentage

SECONDARY OUTCOMES:
Evaluation of periodontium thickness | Before surgery and at the 15-day and 3-month follow-up visits
  Photographs
Evaluation of keratinized tissue width | Before surgery and at the 15-day and 3-month follow-up visits
  Measures using a periodontal probe
Evaluation of the periodontal biotype | Before surgery and at the 15-day, 3-month, 12-months and 24-months follow-up visits
  Maynard and Wilson classification
Surgeon aesthetic evaluation using a visual analogue scale (VAS) scored from 1 to 10 (1=unsatisfactory; 10=very satisfactory). | At the 15-day, 3-month, 12-months and 24-months follow-up visits
  Described at each visit
Patient-reported pain using a visual analogue scale (VAS) scored from 0 to 10 (0=no pain; 10=worse pain). | At the 15-day, 3-month, 12-months and 24-months follow-up visits
  Described at each visit
Patient satisfaction using a visual analogue scale (VAS) scored from 1 to 10 (1=unsatisfactory; 10=very satisfactory). | At the 15-day, 3-month, 12-months and 24-months follow-up visits
  Described at each visit
Device malfunctions-deficiencies: inadequacy of a medical device with respects to its identity, quality, durability, reliability, safety or performance. Device deficiencies include malfunctions, use errors, and inadequate labelling. | During the surgical procedure
  Summarized and listed

CONTACTS AND LOCATIONS:
Overall Officials: Rémy CAHUZAC, Principal Investigator — Cabinet dentaire des chênes, Saint Pierre du Mont, France
Locations (5):
- France (5):
  - Cabinet dentaire Grange Blanche, Lyon
  - Cabinet PISB, Saint-Brieuc
  - CMCT (Centre Médico-Chirurgical de Touraine), Saint-Cyr-sur-Loire
  - Cabinet dentaire des chênes, Saint-Pierre-du-Mont
  - Cabinet dentaire Saint Priest en Jarez, Saint-Priest-en-Jarez

IPD SHARING:
Plan to Share IPD: No